CLINICAL TRIAL: NCT04769739
Title: Comparing Left Colon Mucus Production by Water Versus Saline Infusion During Water Exchange Colonoscopy: a Prospective Randomized Controlled Trial
Brief Title: Dose the Saline Reduce the Mucus Production When Water Exchange Colonoscopy is Used?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: EGH-2021-2
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-04

CONDITIONS: Colon Mucous; Colonoscopy
Keywords: Colonoscopy; Colon Mucus; Water Exchange; Saline
MeSH Terms: interventions — Water; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CO2 insufflation (Active Comparator): Colonoscopy will be performed in the traditional fashion, with minimal insufflation required to aid insertion. Cleaning in the CO2 group will be performed entirely during withdrawal.
  Interventions: Other: CO2
- WE with water (Active Comparator): Residual air in the colon will be removed, water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual decal debris, predominantly during insertion.
  Interventions: Other: Water
- WE with 50% saline (Experimental): Residual air in the colon will be removed, 50% salline (1:1 mixture of saline and water) will be infused to guide insertion through an airless lumen. Infused saline will be removed by suction, along with residual decal debris, predominantly during insertion.
  Interventions: Other: 50% saline
- WE with 25% saline (Experimental): Residual air in the colon will be removed, 25% saline (1:3 mixture of saline and water) will be infused to guide insertion through an airless lumen. Infused saline will be removed by suction, along with residual decal debris, predominantly during insertion.
  Interventions: Other: 25% saline

INTERVENTIONS:
Other: CO2 — using CO2 insufflation to help insertion
  Arms: CO2 insufflation
Other: Water — using water instead of traditional gas to help insertion
  Arms: WE with water
Other: 50% saline — using 50% saline solution instead of traditional gas to help insertion
  Arms: WE with 50% saline
Other: 25% saline — using 25% saline solution instead of traditional gas to help insertion
  Arms: WE with 25% saline

SUMMARY:
This is a study to compare the left colon mucus production between carbon dioxide (CO2) insufflation and water exchange (WE) colonoscopy in patients that require a routine or repeat colonoscopy. There will be four arms in this study: CO2 insufflation (control group 1), WE with water infusion (control group 2), WE with 50% saline infusion (study group 1), and WE with 25% saline infusion (study group 2). The patient will prepare himself/herself for the colonoscopy as per normal instructions and he/she will be given the information for the study at that time so that he/she can make a decision to participate in the study. The WE control group will use sterile water filling during colonoscope insertion. The study method will use saline filling during colonoscopy insertion. This study will confirm if using the saline infusion is a better method in reducing mucus production when WE colonoscopy is used.

DETAILED DESCRIPTION:
This will be a single-site (Evergreen General Hospital, Taoyuan, Taiwan), blinded investigators, prospective randomized controlled trial (RCT). Felix W. Leung (from Sepulveda Ambulatory Care Center, Veterans Affairs Greater Los Angeles Healthcare System, North Hills, CA) will be involved in the study design, data analysis, and report preparation, but not in patient enrollment. Randomization (CO2, WE with water, WE with 50% saline, WE with 25% saline) will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope (in pre-arranged order) will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. This will be a comparison of two different insertion methods with four arms (CO2 insufflation, WE with water, WE with 50% saline, WE with 25% saline) to see which solution used in WE is better in reducing mucus production.

Patients who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Randomization will be stratified by investigators and indication of colonoscopy (screening, surveillance, or positive fecal immunochemical test). All participating patients will receive conscious sedation during the colonoscopic examination. Randomization (prepared by statistics consultant) will be carried out by the method of random permuted block design (based on computer generated random numbers) with variable block of 3 and 6.

Control method: One arm of the study will include colonoscopy with water infusion during insertion as the control method. Residual air in the colon will be removed and sterile water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion. Another arm of the study will include colonoscopy with CO2 insufflation during insertion as an additional control method.

Study method: Two arms of the study will include colonoscopy with saline infusion of different strength, i.e., 50% saline and 25% saline, during insertion. Residual air in the colon will be removed and saline solution will be infused to guide insertion through an airless lumen. Infused saline will be removed by suction, along with residual fecal debris, predominantly during insertion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 20-75 years of age
* Positive screening for Fecal Immunochemical Test (FIT)
* Subjects willing to undergo routine screening and surveillance colonoscopy

Exclusion Criteria:

* Patients who decline to provide informed consent
* Patients known to have colonic obstruction, active inflammatory bowel disease, or active GI bleeding requiring interventions
* Patients known to have prior history of colonic resection
* Patients with genetic colorectal syndromes
* Patients who are scheduled for therapeutic colonoscopy (e.g., hemostasis, removal of large polyp)
* Patients with American Society of Anesthesiology classification of physical status grade 3 or higher

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chiliang Cheng, MD, Principal Investigator — Evergreen General Hospital, Taoyuan, Taiwan
Locations (1):
- Evergreen General Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Rahyel A, McWhinney CD, Parsa N, Lahr RE, Vemulapalli KC, Rex DK. Room temperature water infusion during colonoscopy insertion induces rectosigmoid colon mucus production. Endoscopy. 2020 Dec;52(12):1118-1121. doi: 10.1055/a-1182-5211. Epub 2020 Jun 15. PMID 32458999
- [Background] Anderson JC, Kahi CJ, Sullivan A, MacPhail M, Garcia J, Rex DK. Comparing adenoma and polyp miss rates for total underwater colonoscopy versus standard CO2: a randomized controlled trial using a tandem colonoscopy approach. Gastrointest Endosc. 2019 Mar;89(3):591-598. doi: 10.1016/j.gie.2018.09.046. Epub 2018 Oct 24. PMID 30367879
- [Background] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Derived] Cheng CL, Kuo YL, Liu NJ, Lien JM, Su IC, Tang CP, Hsieh YH, Leung FW. Randomized Trial Comparing Left Colon Mucus Production Using Water vs Saline During Water Exchange Colonoscopy. Clin Transl Gastroenterol. 2023 Jul 1;14(7):e00594. doi: 10.14309/ctg.0000000000000594. PMID 37141104

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Started | 73 | 75 | 76 | 77
Completed | 70 | 75 | 76 | 75
Not Completed | 3 | 0 | 0 | 2
Not completed — Colorectal cancer obstruction | 2 | 0 | 0 | 0
Not completed — Failed cecal intubation | 1 | 0 | 0 | 1
Not completed — Poor bowel preparation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline | Total
Number analyzed (Participants) | 70 | 75 | 76 | 75 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (10.0) | 51.4 (10.7) | 53.0 (11.5) | 52.0 (10.9) | 51.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 43 | 38 | 150
  Male | 33 | 43 | 33 | 37 | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 70 | 75 | 76 | 75 | 296

OUTCOME MEASURES:

1. Primary Outcome: Left Colon Mucus Score
Description: The amount of residual mucus in the left colon (descending colon, sigmoid colon, rectum) is scaled by a mucus score (5-point scale): score 0: no visible mucus; score 1: minimal amounts of clear mucus in thin streaks or strands; score 2: mild opaque mucus in thin strands; score 3: moderate opaque mucus in thicker clumps covering one side of surface; score 4: more opaque mucus in thicker clumps covering more views of lumen.
Time Frame: 2 hours (data collected during colonoscopy procedure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
score on a scale | 0.2 (0.38) | 1.4 (0.84) | 0.5 (0.50) | 0.7 (0.63)

2. Secondary Outcome: Adenoma Detection Rate
Description: The percentage of individuals undergoing a complete screening colonoscopy who have one or more adenomas detected according to the pathology reports.
Time Frame: one week (data analyzed after the pathology results were available)
Measure: Count of Participants; unit: Participants
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
Participants | 35 | 31 | 41 | 35

3. Secondary Outcome: Number of Participants With Cecal Intubation
Description: Number of participants who had a colonoscopy images confirming visualization of ileocecal valve/appendix orifice and the medial wall of the cecum with colonoscope tip touching floor of cecum
Time Frame: 2 hours (data collected during colonoscopy procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
Participants | 70 | 75 | 76 | 75

4. Secondary Outcome: Boston Bowel Preparation Scale Score
Description: Three iindividual segments (right colon, transverse colon, left colon), each with score of 0 to 3 (poor to excellent) will be evlauated separately using the Boston Bowel Preparation Scale. A tota Boston Bowel Preparation Scale score, sum of three-segmental score (range 0-9), will be reported.
Time Frame: 2 hours (data collected during colonoscopy procedure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
score on a scale | 7.0 (0.5) | 7.1 (0.7) | 7.8 (0.7) | 7.6 (0.7)

5. Secondary Outcome: Cecal Intubation Time
Description: Total time from insertion into the anus to arrival in the cecum
Time Frame: 2 hours (data collected during colonoscopy procedure)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
minutes | 10.0 (6.0) | 18.0 (6.2) | 18.4 (7.1) | 18.6 (9.1)

6. Secondary Outcome: Withdrawal Inspection Time
Description: Total inspection time during withdrawal from the cecum to the anus
Time Frame: 2 hours (data collected during colonoscopy procedure)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
Number analyzed (Participants) | 70 | 75 | 76 | 75
minutes | 20.2 (6.4) | 17.1 (5.4) | 17.2 (5.3) | 16.6 (5.4)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | CO2 Insufflation | WE With Water | WE With 50% Saline | WE With 25% Saline
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/75 | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/75 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/70 | 0/75 | 0/76 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT04769739/Prot_SAP_000.pdf